CLINICAL TRIAL: NCT01360528
Title: Zekai Tahir Burak Maternity and Teaching Hospital
Brief Title: Serum Folic Acid Levels in Preterm Infants
Acronym: FALIPI
Status: Completed | Type: Observational
Sponsor: Mehmet Yekta (Other)
Responsible Party: Sponsor-Investigator, Mehmet Yekta, Zekai Tahir Burak Maternity and Teaching Hospital, Zekai Tahir Burak Women's Health Research and Education Hospital
Organization: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Other Study IDs: ztb5326315185
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Very Low Birth Weight Baby
Keywords: Folic acid replacement; Folic acid; Preterm neonate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Extremely low birth weight: Extremely low birth weight under 1000 gram
- Very low birth weight: Between 1000-1500 gram babies
- Low birth weight: Between 1500-2500 gram

SUMMARY:
Therefore preterm infants must need folic acid replacement than term babies.

DETAILED DESCRIPTION:
All babies need to different vitamin supplementation. Especially preterm infants need some vitamin supplements. Folic acid is very important structure of part of cell growing.ın theorically; preterm infants have very rapid cell reproduction capacity than term infants. Therefore preterm infants must need folic acid replacement than term babies. The investigators want to determine preterm infants folic acid levels due to gestational age whether needs folic acid replacement.

ELIGIBILITY:
Inclusion Criteria:

-All preterm infants

Exclusion Criteria:

-Major congenital anomaly

Ages: 24 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Extremely low birth weight, Very low birth weight, Low birth weight
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Neonatology Unit, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Oncel MY, Calisici E, Ozdemir R, Yurttutan S, Erdeve O, Karahan S, Dilmen U. Is folic acid supplementation really necessary in preterm infants </= 32 weeks of gestation? J Pediatr Gastroenterol Nutr. 2014 Feb;58(2):188-92. doi: 10.1097/MPG.0000000000000181. PMID 24051483